CLINICAL TRIAL: NCT02161549
Title: Evaluation of the Motus Gl CleanUp System During Screening Colonoscopy
Status: Completed | Type: Observational
Sponsor: Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-MCU-SP-1211
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-03

CONDITIONS: CRC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colonoscopy with MotusGi CleanUp System Rev 1.0: subjects indicated for colonoscopy procedure with CleanUp System Rev 1.0 , enrolled under protocol Rev 1.0
  Interventions: Device: Motus Gl CleanUp System
- Colonoscopy with MotusGi CleanUp System Rev 1.5: subjects indicated for colonoscopy procedure with CleanUp System Rev 1.5 , enrolled under protocol Rev 2.0
  Interventions: Device: Motus Gl CleanUp System

INTERVENTIONS:
Device: Motus Gl CleanUp System

SUMMARY:
Motus Gl is developing a single-use device that attaches to a standard colonoscope, thereby integrating colon cleansing, screening and treatment into one procedure.

The device creates turbulence within the colon using water jets. The colon's fecal fluids are evacuated by the system.

DETAILED DESCRIPTION:
63 eligible subjects who are allocated for a diagnostic screening colonoscopy were enrolled in the study. The assignment of the level of the bowel preparation agent was according to the physician decision. Following preparation, enrolled subjects were intubated and cleansed using a standard colonoscope with the Motus GI CleanUp device attached to it. At the end of the procedure, subjects were followed through discharge and at 48 hours post procedure for occurrence of adverse events.

40 subjects were enrolled under protocol Rev 1.0 used Motus GI CleanUp System Rev 1.0 31 subjects were enrolled under protocol Rev 2 used Motus GI CleanUp System Rev 1.5, due to improvement made to the study device including the following:

1. One head that irrigates and evacuates instead of two heads
2. Elimination of the grinding mechanism and the motor to reduce the pipes' diameters while keeping the same flow rate.
3. System adjustment to the above changes including updated software version.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in the age range of 50-69 years
* Subjects who are considered for routine screening colonoscopy
* Subjects with BMI within the range of 18.5-30
* Subject is willing to sign informed consent form

Exclusion Criteria:

* History of G diseases or history of Colorectal cancer (personal or family)
* Previous major abdominal surgeries
* Medical status ASA grater or equal to 3
* Acute Gl symptoms, such as bleeding, unexplained weight loss, inflammatory bowel disease (lBD).
* Patients taking anticoagulants (e.g., Coumadin, Heparin, Clopidrogrel)
* Life-threatening condition
* Subjects who are unable or unwilling to cooperate with study procedures
* Severe Diverticula

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects indicate for standard colonoscopy procedure (i.e., screening, diagnostic , surveillance)
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica San Rafael, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was done in two phases:
  Phase 1- under protocol Rev 1.0 used MotusGi CleanUp System Rev 1.0 , study period Aug- Jan 2012. 40 subjects enrolled.
  Phase 2- under protocol Rev 2.0 used MotusGi CleanUp System Rev 1.5 , study period Jul-Oct 2013.31 subjects enrolled.
Groups:
- Colonoscopy With MotusGi CleanUp System Rev 1.0: subjects indicated for colonoscopy procedure with CleanUp System Rev 1.0 , enrolled under protocol Rev 1.0
  Motus Gl CleanUp System
- Colonoscopy With MotusGi CleanUp System Rev 1.5: subjects indicated for colonoscopy procedure with CleanUp System Rev 1.5 , enrolled under protocol Rev 2.0
  Motus Gl CleanUp System
Period: Overall Study
Arm/Group | Colonoscopy With MotusGi CleanUp System Rev 1.0 | Colonoscopy With MotusGi CleanUp System Rev 1.5
Started | 40 | 31
Completed | 34 | 29
Not Completed | 6 | 2
Not completed — Physician Decision | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colonoscopy With MotusGi CleanUp System Rev 1.0 | Colonoscopy With MotusGi CleanUp System Rev 1.5 | Total
Number analyzed (Participants) | 34 | 29 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (3.8) | 53 (4.1) | 54 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 21 | 15 | 36

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of Boston Bowel Preparation Scale (BBPS) Index Prior and After the Use of MotusGI CleanUp System
Description: Human colon has 3 segments and each segment can be scored 0 (unprepared colon) - 3 (clean colon). average of all colon segments BBPS score after the use of MotusGI CleanUp System
Time Frame: during colonoscopy procedure after cleansing with CleanUp System
Population: the mean and standard deviation of the average score after cleansing the colon using the Motus CleanUp System
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Colonoscopy With MotusGi CleanUp System Rev 1.0 | Colonoscopy With MotusGi CleanUp System Rev 1.5
Number analyzed (Participants) | 34 | 29
units on a scale | 2.9 (0.4) | 2.9 (0.2)

ADVERSE EVENTS:
Arm/Group | Colonoscopy With MotusGi CleanUp System Rev 1.0 | Colonoscopy With MotusGi CleanUp System Rev 1.5
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/31
Other Adverse Events (participants affected / at risk) | 17/40 | 17/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colonoscopy With MotusGi CleanUp System Rev 1.0 (N=40) | Colonoscopy With MotusGi CleanUp System Rev 1.5 (N=31)
Erosion (Gastrointestinal disorders) | 5 (7) | 13 (13) — mild erosion probably related to colonoscopy procedure resolved without clinical intervention
Hematoma (Gastrointestinal disorders) | 5 (11) | 7 (8) — mild Hematoma resolved without clinical intervention
Vesicles (Gastrointestinal disorders) | 3 (3) | 0 (0) — mild
Laceration (Gastrointestinal disorders) | 0 (0) | 6 (6) — 5 mild and 1 moderate lacerations resolved without clinical intervention
Papules (Gastrointestinal disorders) | 4 (5) | 0 (0) — mild Papules resolved without clinical intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No